CLINICAL TRIAL: NCT01091389
Title: A Randomized Single Center Study to Prospectively Investigate the Effect of Ablation of the Autonomic Ganglia in Addition to Minimally Invasive Surgical Isolation of Pulmonary Veins in Patients With Atrial Fibrillation
Brief Title: Atrial Fibrillation Ablation and Autonomic Modulation Via Thorascopic Surgery
Acronym: AFACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Principal Investigator, J.R. de Groot, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL30199.018.10
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Totally Thoracoscopic PV isolation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Maze Procedure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GP ablation (Experimental): Thoracoscopic PV isolation with GP ablation
  Interventions: Procedure: Totally Thoracoscopic PV isolation
- No GP ablation (Experimental): Thoracoscopic PV isolation with no GP ablation
  Interventions: Procedure: Totally Thoracoscopic PV isolation

INTERVENTIONS:
Procedure: Totally Thoracoscopic PV isolation — Surgery is performed through three ports bilaterally in the intercostal spaces. PVI is performed with a bipolar radiofrequency clamp and confirmed with a custom made multi-electrode probe with closely spaced (1mm) electrode terminals. Additional left atrial ablation lines are created and conduction block is verified in patients with persistent and permanent AF.
  Other Names: Mini-Maze; VATS-PVI

SUMMARY:
This study aims at investigating the role of autonomic modulation of AF. Therefore, totally thoracoscopic PV isolation with additional ablation of ganglionated plexi (GP) will be studied against PV isolation alone. Two groups of patients (paroxysmal AF with or without structural heart disease and persistent AF with or without heart disease) of 110 patients each will be studied.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common chronic arrhythmia in man. Its treatment consists of control of ventricular rate or attempts to restore sinus rhythm. For symptomatic patients who fail on anti arrhythmic drugs, isolation of the pulmonary veins (PV), with additional linear left atrial lesions when appropriate, can cure AF. At least in some, but probably in many patients, the autonomous nervous system plays a pivotal role in the initiation and perpetuation of AF. The autonomic ganglia, or ganglionated plexi (GP) are located within the epicardial fat pads of the left atrium. This study aims at investigating the additional value of ablation of those GPs in addition to totally thoracoscopic PV isolation.

Objective of the study:

This study aims at investigating the role of autonomic modulation of AF. Therefore, totally thoracoscopic PV isolation with additional ablation of ganglionated plexi (GP) will be studied against PV isolation alone. Two groups of patients (paroxysmal AF with or without structural heart disease and persistent AF with or without heart disease) of 110 patients each will be studied.

Study design:

This is a single center, randomized single blinded study

Study population:

Any patient with an indication for non-pharmacological treatment of symptomatic paroxysmal or persistent AF can enter the study. An indication for non-pharmacological treatment exists when patients are symptomatic and have failed on at least one anti-arrhythmic drug. Symptoms of AF include, but are not limited to palpitations, reduced exercise capacity, exertional dyspnea, and fatigue. Failure of anti-arrhythmic therapy is defined as 1) recurrence of AF despite the use of an anti-arrhythmic drug in a clinical efficacious dosing or 2) adverse effects of medication that is not acceptable to the patient.

Intervention (if applicable):

In patients randomized to additional GP ablation, the following procedures will be carried out during the totally thoracoscopic procedure in addition to the PV isolation (and extended lesion set when appropriate): The left atrial autonomic GPs are localized within the epicardial fat pads and subsequently ablated with radiofrequency current delivered through an ablation probe (AtriCure Isolator™ Transpolar™ pen).

ELIGIBILITY:
Inclusion Criteria:

* Age is between 18 and 80 years
* AF is symptomatic, paroxysmal or persistent (hence not long standing persistent)
* In case of persistent AF, successful cardioversion within the last 12 months (cardioversion will be considered failed if AF recurs within 48 hours)
* AF was documented on ECG, Holter or pacemaker electrogram at least once in the 6 months preceding presentation
* At least one class I or III antiarrhythmic drug in standard dosage has failed or is not tolerated
* Legally competent and willing and able to sign informed consent
* Willing and able to adhere to the follow up visit protocol
* Life expectancy of ≥2 years

Exclusion Criteria:

* Prior catheter ablation for AF within the preceding 4 months
* Refusal to take antiarrhythmic medication
* Myocardial infarction (defined as CKMB> twice upper limit of normal) within the preceding 2 months
* NYHA class IV/IV heart failure symptoms, or class II-III with a recent decompensation requiring hospitalization or left ventricular ejection fraction<35% (unless related to or aggravated by AF).
* Cerebrovascular accident (defined as any sudden neurological deficit lasting longer than 24 hours, with or without pathological changes on the CT cerebrum) with the preceding 6 months
* Known and documented carotid stenosis>80%
* Planned cardiac surgery for other purposes than AF (alone)
* Evidence of active infection (as evidenced by increased white blood cell count, elevated CRP level or fever >38,5 °C)
* Unable to undergo TEE
* Pregnancy or of childbearing potential without adequate contraception
* Requirement of antiarrhythmic medication for ventricular arrhythmias
* Presence of intracardiac mass or thrombus (Discovery of any thrombus or intracardiac mass after signing of the informed consent will result in withdrawal of the patient from the study)
* Co-morbid condition that possesses undue risk of general anesthesia or port access cardiac surgery (in the opinion of the investigator)
* History of previous radiation therapy on the thorax
* Circumstances that prevent follow-up (no permanent home or address, transient, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-03; Primary Completion 2015-02-23 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is freedom of AF after one year after the procedure without the use of antiarrhythmic drugs. | One year
  The primary endpoint of the study is freedom of AF after one year after the procedure without the use of antiarrhythmic drugs. Freedom of AF is defined as the absence of documentation of AF on serial Holter recordings during follow up and on ECGs recorded outside the scope of the study. One single episode of <30 minutes is allowed. Patients complaints about palpitations without the documentation of AF is allowed.

SECONDARY OUTCOMES:
Freedom of AF after two years after the procedure without the use of any antiarrhythmic drug | Two Years
  Freedom of AF after two years after the procedure without the use of any antiarrhythmic drug. Definition of freedom of AF as above.
Quality of life | One Year
  Improvement of functional status as measured by the RAND 36 quality of life questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: J.R. De Groot, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands

REFERENCES:
- [Result] Driessen AHG, Berger WR, Krul SPJ, van den Berg NWE, Neefs J, Piersma FR, Chan Pin Yin DRPP, de Jong JSSG, van Boven WP, de Groot JR. Ganglion Plexus Ablation in Advanced Atrial Fibrillation: The AFACT Study. J Am Coll Cardiol. 2016 Sep 13;68(11):1155-1165. doi: 10.1016/j.jacc.2016.06.036. PMID 27609676
- [Derived] Wesselink R, Neefs J, van den Berg NWE, Meulendijks ER, Terpstra MM, Kawasaki M, Nariswari FA, Piersma FR, van Boven WJP, Driessen AHG, de Groot JR. Does left atrial epicardial conduction time reflect atrial fibrosis and the risk of atrial fibrillation recurrence after thoracoscopic ablation? Post hoc analysis of the AFACT trial. BMJ Open. 2022 Mar 9;12(3):e056829. doi: 10.1136/bmjopen-2021-056829. PMID 35264365
- [Derived] Reyat JS, Chua W, Cardoso VR, Witten A, Kastner PM, Kabir SN, Sinner MF, Wesselink R, Holmes AP, Pavlovic D, Stoll M, Kaab S, Gkoutos GV, de Groot JR, Kirchhof P, Fabritz L. Reduced left atrial cardiomyocyte PITX2 and elevated circulating BMP10 predict atrial fibrillation after ablation. JCI Insight. 2020 Aug 20;5(16):e139179. doi: 10.1172/jci.insight.139179. PMID 32814717
- [Derived] Berger WR, Neefs J, van den Berg NWE, Krul SPJ, van Praag EM, Piersma FR, de Jong JSSG, van Boven WP, Driessen AHG, de Groot JR. Additional Ganglion Plexus Ablation During Thoracoscopic Surgical Ablation of Advanced Atrial Fibrillation: Intermediate Follow-Up of the AFACT Study. JACC Clin Electrophysiol. 2019 Mar;5(3):343-353. doi: 10.1016/j.jacep.2018.10.008. Epub 2018 Nov 28. PMID 30898238